CLINICAL TRIAL: NCT06358989
Title: Association Between Triglycerides Glucose Ratio With HOMA -IR as Indicators of Insulin Resistance in Obese Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Esmat Mohamed Kotb, Resident doctor, Assiut University
Other Study IDs: Insulin resistance
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: HOMA IR — Homa ir

SUMMARY:
The aim of the present study was to investigate the correlation between the triglyceride/glucose index (TyG index) and homeostasic model assessment of insulin resistance (HOMA-IR) to predict insulin resistance (IR) in obese adults

DETAILED DESCRIPTION:
Obesity is a chronic disease that has an increasing prevalence in both developed and developing countries and affects adults and children[1] Obesity is an important risk factor for the development of some chronic diseases such as insulin resistance, hypertension, and type 2 diabetes [2]

. Insulin sensitivity is inversely related to body mass index and body fat. Insulin resistance can be defined as impairment of the normal biological response to both endogenous and exogenous insulin. One of the primary defects underlying the development of type 2 diabetes is thought to be insulin resistance. So, it is present in 85% of these patients with Type 2 DM. It is also related to the pathogenesis of many illnesses which includes coronary heart disease, and hypertension[3] Early detection of insulin resistance (IR) is important to prevent the development of cardiometabolic diseases such as Type 2 Diabetes Mellitus, metabolic syndrome, and coronary heart disease. The Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) index, which has high sensitivity and specificity, has been shown to be more useful in estimating the risk of insulin resistance, instead of more invasive, complex, and expensive direct tests such as pancreatic suppression test and hyperinsulinemic-euglycemic glucose clamp technique [4] HOMA-IR is an approved method for evaluating insulin resistance using fasting glucose and insulin levels and is widely used in clinical practice [5].

Triglyceride glucose (TyG) index is a novel marker, which has been demonstrated to have a high sensitivity and specificity in identifying insulin resistance [6].

Recently, the use of the triglyceride glucose (TyG) index, a product of fasting glucose and triglyceride are more easily accessible assessment tools both at the outpatient clinics and at the community level, and are low cost [7].

ELIGIBILITY:
Inclusion Criteria:

* Any obese adult (18 years or older) with BMI greater than or equal 30 of both sexes admitted to assiut unversity hospitals and clinics

Exclusion Criteria:

* Cases <18 years old
* Cases with BMI < 30
* Adult with endocrine abnormatilies under treatment for DM ,hypertension , dyslipidemia

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any obese adult (18 years or older) with BMI greater than or equal 30 of both sexes admitted to assiut unversity hospitals and clinics
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Association between triglycerides glucose ratio with HOMA -IR as indicators of insulin resistance in obese adults | Baseline
  The study is to investigate the usability of the Ty-G index as an indicator of insulin resistance in obese adults according to its correlation with HOMA-IR

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Bittner V, Johnson BD, Zineh I, Rogers WJ, Vido D, Marroquin OC, Bairey-Merz CN, Sopko G. The triglyceride/high-density lipoprotein cholesterol ratio predicts all-cause mortality in women with suspected myocardial ischemia: a report from the Women's Ischemia Syndrome Evaluation (WISE). Am Heart J. 2009 Mar;157(3):548-55. doi: 10.1016/j.ahj.2008.11.014. PMID 19249427